CLINICAL TRIAL: NCT01545115
Title: Study of the Environmental Factors Modulating Children Immune Response in Northern Senegal
Acronym: AnoPalAnoVac
Status: Completed | Type: Observational
Sponsor: Biomedical Research Center EPLS (Other)
Collaborators: Institut Pasteur de Lille (Other); Institut de Recherche pour le Developpement, Senegal (Other); Institut de Recherche pour le Developpement (Other Government); University of Lille Nord de France (Other); Région Nord-Pas de Calais, France (Other); Centre d'Infection et d'Immunité de Lille (Other); Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: EPLS08-JBS
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Whooping Cough; Malaria; Malnutrition
Keywords: Children; Immunity; Sub-Saharan; Pertussis; Malaria; Nutrition; antibodies
MeSH Terms: conditions — Whooping Cough; Malaria; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera, culture supernatants
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Longitudinal survey in Northern Senegal to investigate the environmental factors modulating the immune response to childhood vaccines and to malaria.

A cohort of 410 children aged 1 to 10 from 5 villages of the Senegal River Valley(Podor District) was followed-up for 18 months. During that period, 5 visits have been made to the villages to assess the immunological and nutritional status of the children.

DETAILED DESCRIPTION:
Longitudinal survey in Northern Senegal to investigate the environmental factors modulating the immune response to childhood vaccines and to malaria.

A cohort of 410 children aged 1 to 10 from 5 villages of the Senegal River Valley(Podor District) was followed-up for 18 months. During that period, 5 visits have been made to the villages to assess the immunological and nutritional status of the children (T1 (October 2008), T2 (January 2009), T3 (June 2009), T4 (October 2009) and T5 (January 2010)).

The project was approved by the National Ethics Committee of Senegal. Written individual informed consent was obtained from each participant's parent or legal guardian at the beginning of the survey, and at each visit child's and parent's approval was sought orally.

Capillary blood was collected from the finger tip of each child, using sterile single-use material.

Body temperature was measured by means of auricular thermometer at all visits. Anthropomorphic data were collected at visits T2, T3, T4 and T5.

A Hemocue photometer (HemoCue AB, Ängelholm, Sweden) was used to determine haemoglobin concentration on a blood drop at visits T3, T4 and T5.

At each visit, a questionnaire was filled in for every child. Information was collected on the date of birth family membership to asses if siblings or children living in the same house were in the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 1 and 10 years

Exclusion Criteria:

* Fever (body temperature superior to 38.5 °C)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Residents of 5 villages from the Senegal Valley River, belonging to the Podor District in Saint-Louis Region in Northern Senegal.
  Agniam (16°32'N-14°48'W; total population (TP): 989; several temporary ponds, traditional housing, irrigated crops) Fanaye Diery (16°32'N-15°13'W; TP: 6781; animal husbandry, irrigated crops, some urbanized habitat) Niandane (16°35'N-14°59'W; TP: 5100; Rice and banana farming, irrigated crops, some urbanized habitat) Ndiayène Pendao (16°30'N- 15°03'W; TP: 2734; animal husbandry, Savannah surroundings) Guédé Village (16°33'N-14°48'W; TP:3005; Traditional housing, irrigated crops)
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Remoué, PhD, Study Chair — Biomedical Research Center EPLS; Emmanuel Hermann, PhD A. Pr., Study Director — Biomedical Research Center; Jean Biram Sarr, PhD, Principal Investigator — Biomedical Research Center EPLS; Lobna Gaayeb, VetMed, Principal Investigator — Biomedical Research Center EPLS
Locations (1):
- Biomedical Research Center EPLS, Saint-Louis, Saint-Louis, Senegal

REFERENCES:
- [Background] Ndiath MO, Sarr JB, Gaayeb L, Mazenot C, Sougoufara S, Konate L, Remoue F, Hermann E, Trape JF, Riveau G, Sokhna C. Low and seasonal malaria transmission in the middle Senegal River basin: identification and characteristics of Anopheles vectors. Parasit Vectors. 2012 Jan 23;5:21. doi: 10.1186/1756-3305-5-21. PMID 22269038
- [Derived] Gaayeb L, Pincon C, Cames C, Sarr JB, Seck M, Schacht AM, Remoue F, Hermann E, Riveau G. Immune response to Bordetella pertussis is associated with season and undernutrition in Senegalese children. Vaccine. 2014 Jun 5;32(27):3431-7. doi: 10.1016/j.vaccine.2014.03.086. Epub 2014 Apr 14. PMID 24726248
- See also: EPLS website — http://www.espoir-sante.org